CLINICAL TRIAL: NCT03958643
Title: Best Noninvasive Predictor of Renal Function in Assessing Adult Sickle Nephropathy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190100; 19-H-0100
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01-13

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Nephropathy; Iothalamate; Cystatin-C; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: In a population of adult patients with SCD we will comprehensively evaluate renal function.

SUMMARY:
Background:

Sickle cell disease is a common inherited blood disorder. Kidney disease is a major cause of problems in people with sickle cell disease. In order to identify kidney problems early and stop the progression of kidney disease, doctors need the most accurate tests to check kidney function. Researchers hope to understand more about how to test for kidney disease in people with sickle cell disease.

Objective:

To determine which of two different lab tests is the best to measure kidney function in adults with sickle cell disease.

Eligibility:

People 18 years and older who have sickle cell disease

Design:

Participants will be screened with a medical history and blood tests.

Participants will have up to 3 visits.

Participants will collect their urine in a special container over 24 hours.

At the first visit, participants will have blood tests. They will bring their container of urine to the visit. They will have an iothalamate test. For the test, they will get a catheter: a small tube will be inserted into a vein. A special contract agent will be injected into the vein. Blood will be collected over the next 4 hours to test kidney function.

Participants will return the next day for a second visit. They will have blood tests. They will have an MRI. For the MRI, they will like on a table that slides into a machine that takes pictures of the kidneys. They may have the MRI in a third visit.

...

DETAILED DESCRIPTION:
The characteristic sickling of red blood cells in hypoxic conditions is the root cause of pathology in sickle cell disease (SCD). When this sickling occurs in the renal microvasculature, and is compounded by chronic vasculopathy related to hemolysis, the result is local infarction, ischemic injury, and interstitial fibrosis. The kidney damage begins in early childhood and is cumulative over time, resulting in sickle cell nephropathy (SCN). Creatinine clearance remains the most commonly used method to evaluate renal function in SCD patients although serum creatinine generally over-estimates the GFR in SCD. Cystatin-C (Cys-C) is freely filtered. Unlike creatinine, it is not secreted by the tubules. Its serum levels correlate with GFR in adults with various kidney diseases as well as in pediatric and adult SCD populations as compared with creatinine-based assessments.

This study seeks to evaluate whether Cys-C is a better noninvasive measure of renal function in the adult sickle cell population than creatinine. Further, this work will elucidate the ability of other markers, including beta 2-microglobulin (beta 2M) and endothelin-1 (ET-1), to predict sickle nephropathy. Finally, renal imaging by MRI will be performed and correlated with measured GFR and renal function markers. The results of this study could help alter clinical practice and thereby ensure the most accurate non-invasive assessment of kidney function by substantiating the role of Cys-C, beta 2M and ET-1 in adults with SCD. Finally, the descriptive analysis including measured GFR with renal MRI, novel biomarkers, markers of hemolysis, and analysis of urinary protein secretion will contribute to a better understanding of the pathophysiology of SCN.

ELIGIBILITY:
* INCLUSION CRITERIA:

Known diagnosis of Sickle Cell Anemia (Hb SS or HbS-beta0-thal) >=18 years of age

Willingness and capacity to provide written informed consent

EXCLUSION CRITERIA:

Pregnancy

Uncontrolled/poorly controlled hypertension

Diabetes

Dialysis

GFR <30 ml/min/1.73m2

HIV positive

HepatitisC

Hepatitis B

Prior transplantation

Uncontrolled infection or acute illness

Chronic inflammatory disease (e.g. lupus, multiple sclerosis, rheumatoid arthritis)

Allergy to iodine or iodinated contrast solutions

Hydroxyurea initiation or dose adjustment <2mo prior

Initiation of chronic transfusion therapy <2mo prior

Antihypertensive medication initiation or dose adjustment <1mo prior

Pain crisis in preceding 4weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be open to all eligible subjects based on inclusion and exclusion criteria and who provide informed consent. No patient will be excluded from participation based on gender, race, or ethnicity. Patients may self-refer, be recruited through the NIH office of recruitment, and may include patients participating on NIH Clinical Center Protocols, and NIH employees.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Determine whether serum cystatin C or serum creatinine-based GFR methods better estimate renal function in the adult sickle cell population | 2 years
  In a population of patients with sickle cell anemia (including HbSS, HbS-0 thalassemia), who are age 18 and above, we will comprehensively evaluate renal function with the following primary objective:-determine whether serum cystatin C or serum creatinine- based GFR methods better estimate renal function in the adult sickle cell population

SECONDARY OUTCOMES:
Determine whether endothelin-1 or beta-2 microglobulin correlates with measured GFR (mGFR) | 2 years
  Determine whether endothelin-1 or beta-2 microglobulin correlates with measured GFR (mGFR)-establish potential correlation between mGFR, endothelin-1, or beta-2 microglobulin and renal blood flow-characterize the proteinuria associated with sickle cell disease-characterize kidney anatomy in patients with sickle cell disease-ascertain if markers of hemolysis are associated with mGFR or renal iron deposition-quantify renal iron burden in sickle cell disease

CONTACTS AND LOCATIONS:
Overall Officials: Courtney F Joseph, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-H-0100.html

DOCUMENTS (1):
  • Informed Consent Form (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT03958643/ICF_000.pdf